CLINICAL TRIAL: NCT01640041
Title: Feasibility Study for Enhancing Gait Following Stroke With Implanted Microstimulators
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Alfred E. Mann Foundation for Scientific Research (Other)
Collaborators: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: AMF-CP-0004; GO70151
Record Dates: First submitted 2011-06-22; First posted 2012-07-13 (Estimated); Last update posted 2017-01-25 (Estimated); Status verified 2012-07

CONDITIONS: Hemiparesis
MeSH Terms: conditions — Paresis | interventions — Drug Delivery Systems

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Implanted (Experimental): All participants.
  Interventions: Device: Radio-frequency Microstiumulator

INTERVENTIONS:
Device: Radio-frequency Microstiumulator — All participants will receive leg implants and will be trained first in the clinical and subsequently perform stimulation-assisted exercises in the home - for an overall duration of 6 months post-implant. Subsequently, exercise programs will continue without stimulation. Patient condition will be assessed at 9, 12 and 24 months post-implant.
  Other Names: The specific device name is the Radio Frequency Microstiumlator (RFM) System.

SUMMARY:
The purpose of this study is to test an innovative, advanced FNS microstimulator technology developed by the Alfred Mann Foundation (Santa Clarita, CA) called, the Radio Frequency Microstimulation (RFM) Gait System that promises to provide FNS training for restoration of functional gait components in a manner at least as efficacious as current investigational FNS systems. The design features of the RFM Gait System are intended to address the problems with the current FNS systems. The RFM implant devices are small enough to be inserted using only a 5 mm incision[3]. Because both the electrode (anode and cathode) are contained within the microstimulator, there are no lead wires traversing the skin, joints, or torso/limb junctures. Individual RFMs can be inserted at the motor points and nerves of each of the paretic muscles in the involved limb and coordinated using radio frequency technology.

DETAILED DESCRIPTION:
The primary objective (Aim I) of this study is to evaluate whether the RFM Gait System can restore the capability to perform the components of gait required for safe, functional walking, for patients in the chronic phase after stroke (> 12 months). We will assess the treatment provided by the RFM system at the Cleveland VA compared to the FNS percutaneous Schreiner electrodes and custom-designed controller previously investigated by the investigators.

The similarities between the RFM-based and percutaneous FNS systems will be assessed using six gait components required for the execution of functional, safe gait, which are lower limb strength, coordination, an index of walking endurance, muscle tone, walking speed, and quality of life.

The secondary objective of this study is to test the technological performance and safety of the RFM Gait System. Measures of technology performance and safety include implantation time; anchoring capability at the motor point of the muscle; reliability of the RFMs during use; reliability of electrical performance of the system; comfort of the system (with stimulation off); comfort of the electrical stimulus.

ELIGIBILITY:
Inclusion Criteria:

1. Cognition intact to give valid informed consent to participate.
2. Sufficient endurance to participate in rehabilitation sessions.
3. Ability to follow 2 stage commands, in English.
4. Medically stable.
5. Age > 21 years.
6. Impaired ambulation as follows: inability to flex the knee and ankle in the sagittal plane, in a normal manner so the foot clears the floor, inability to control normal knee angle during single limb weight bearing during stance phase .
7. Minimum trace (Manual Muscle Test score of 1) contraction of hip, knee, and ankle flexors and extensors under volitional control.
8. Passive range of motion at hip, knee, ankle normal gait kinematics.
9. Five degrees (5°) of motion for knee and ankle flexors and extensors produced by muscle stimulation achieved non-invasively with electrical stimulation applied to the skin surface.
10. At least 12 months post stroke.
11. Ability to understand the informed consent form in English.
12. Thigh and lower leg circumference and length ≤ 50th percentile of standard U.S. population morphology measures.*
13. Participants should be able to walk and keep balance without physical assistance
14. Response to Surface Stimulation at a trace for tibialis anterior and peronous longus.
15. Subject with unilateral defects

Exclusion Criteria:

1. Acute or progressive cardiac, renal, respiratory, neurological disorders or malignancy.
2. Active psychiatric diagnosis or psychological condition, or active drug/alcohol abuse.
3. Lower motor neuron damage or radiculopathy.
4. More than one stroke.
5. Allergy or contraindication to the anesthesia, Versed, (or comparable substitute).

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2008-05; Primary Completion 2009-12 (Actual); Study Completion 2010-01 (Actual)

PRIMARY OUTCOMES:
Change from baseline to Month 24 of swing phase gait components and knee control during stance phase with 6 gait components. | 24 months
  The six gait components listed below:
  1. Ankle plantar-flexion at Heel Strike
  2. Ankle Dorsiflexion during Peak Swing
  3. Knee Flexion at Toe Off
  4. Knee Flexion Peak Swing
  5. Knee Extension at Heel Strike
  6. Knee Flexion at Mid Stance

SECONDARY OUTCOMES:
Change from baseline to Month 24, without stimulation, of four scales and two QOL questionnaires. | 24 months
  The four scales are:Six Minute Walk Test, Manual Muscle Test, Fugl-Meyer Coordination Scale, and the Ashworth Scale.
  The two QOL questionnaires are: Craig Handicap Assessment & Reporting Technique (CHART) and Stroke Impact Scale (SIS):

CONTACTS AND LOCATIONS:
Overall Officials: Janis J Daly, PhD, MSPT, Principal Investigator — Cleveland VA Medical Center; Robert Ruff, MD, PhD, Principal Investigator — Cleveland VA Medical Center
Locations (1):
- VA Medical Center, Cleveland, Ohio, United States

REFERENCES:
- [Background] Daly JJ, Roenigk K, Holcomb J, Rogers JM, Butler K, Gansen J, McCabe J, Fredrickson E, Marsolais EB, Ruff RL. A randomized controlled trial of functional neuromuscular stimulation in chronic stroke subjects. Stroke. 2006 Jan;37(1):172-8. doi: 10.1161/01.STR.0000195129.95220.77. Epub 2005 Dec 1. PMID 16322492
- [Background] Daly JJ, Ruff RL. Feasibility of combining multi-channel functional neuromuscular stimulation with weight-supported treadmill training. J Neurol Sci. 2004 Oct 15;225(1-2):105-15. doi: 10.1016/j.jns.2004.07.006. PMID 15465093
- [Background] Daly JJ, Kollar K, Debogorski AA, Strasshofer B, Marsolais EB, Scheiner A, Snyder S, Ruff RL. Performance of an intramuscular electrode during functional neuromuscular stimulation for gait training post stroke. J Rehabil Res Dev. 2001 Sep-Oct;38(5):513-26. PMID 11732829